CLINICAL TRIAL: NCT01990586
Title: An Open Label, Randomised, 2-Period, 2-Treatment, 2-Sequence, Crossover, Single-Dose Bioequivalence Study of Rabeprazole Sodium Delayed Release Tablets 20 mg (Test, Torrent Pharmaceuticals Limited., India) Versus Aciphex® (Rabeprazole Sodium) Delayed Release Tablets 20 mg (Reference, Eisai Inc., USA) in Healthy Human Volunteers Under Fed Condition.
Brief Title: Bioequivalence Study of Torrent Pharmaceutical Ltd.'s Rabeprazole Sodium Delayed Release Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PK-10-067
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Healthy
MeSH Terms: interventions — Rabeprazole; Tablets, Enteric-Coated

INTERVENTIONS:
Drug: Rabeprazole sodium 20 mg Delayed Release tablet

SUMMARY:
Objective:

Primary objective of the present study was to compare the single dose bioavailability of Torrent's Rabeprazole Sodium Delayed Release Tablets 20 mg and Aciphex® Delayed Release Tablets 20 mg (Reference, Eisai Inc., USA). Dosing periods were separated by a washout period during fed study.

Study Design:

Open-Label, Randomised, two Period, two treatment, Crossover, Single-Dose Bioequivalence Study

ELIGIBILITY:
Inclusion Criteria:

* Healthy male human volunteers within the age range of 18 to 50 years
* A body mass index within 18-25 Kg/m2
* Given written informed consent to participate in the study
* Absence Of disease markers of HIV 1& 2, hepatitis B & C virus and RPR.
* Absence of significant disease or clinically' significant abnormal laboratory values on laboratory evaluation, medical history and medical examination during the screening
* A normal 12 lead ECG.
* A normal chest X-ray (FA view)
* Comprehension of the nature and purpose'of the study and compliance with the requirement of the entire protocol
* No history or no evidence of hypersensitivity to rabeprazole substituted benzimidazoles or to any component of the formulation
* No history of Anaphylaxis arid Angioedema
* No history or presence of gastric malignancy
* No history of significant systemic diseases
* No history of psychiatric disorders
* No history of addiction to any recreational drug or drug dependence
* No donation of blood(one unit or 350 mL) within 90 days prior to study check-in
* No participation in any clinical study within the last 90 days
* No receipt of any prescription drugs or over-the-counter drugs (e.g.: Cold preparations, and antacid preparations' vitamins and natural products used for therapeutic benefits), within two weeks prior to study check-in
* No history of dehydration from diarrhea, vomiting or any other reason within a period of 24.0 hours prior to study check-in
* No family history of neurological disorders
* Not consumed alcohol and xanthin containing food and beverages, (chocolates, tea,coffee or cola drinks) cigarettes and tobacco products for at least 48.0 hours prior to study check-in for each period.
* Negative results for drugs of abuse (Benzodiazepines, Cocaines, Opioids, Amphetamines, Cannabinoids and Barbiturates) in urine during the day of study check-in of each period
* Not consumed grapefruit(mosumbi/sweet lime) juice within the 48.0 hours prior to study check-in
* Negative alcohol breath analysis during the study check-in of each period

Exclusion Criteria:

* History of seizures
* Received pharmacological agents known to significantly induce or inhibit drug metabolizing enzymes within 14 days of the start of the study
* History of alcohol consumption for more than two units/day (1 unit=30 mL of spirit/or 1 pint of beer), or having consumed alcohol within 48.0 hours prior to check-in
* High caffeine (more than 5 cups of coffee or tea/day) or tobacco (mote than 9 cigarettes/beedies/cigars per day) consumption
* History of difficulty with donating blood or difficulty in accessibility of veins
* An unusual or abnormal diet for whatever reason e.g. because of fasting due to religious reasons

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Primary Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
bioequivalence based on Composite of Pharmacokinetics | plasma samples were obtained from blood drawn at Pre-dose and 0.5, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 4.50, 5.00, 5.50, 6.00, 6.50, 7.00, 8.00, 10.00, 12.00, 14.00, 18.00 and 24.00 hours after dose administration
  bioequivalence; 90% geometric confidence interval of the ratio of least-squares means of the test to reference product should be within 80.00% - 125.00% for AUC-unf, AUCo-t and Cmax.

CONTACTS AND LOCATIONS:
Locations (1):
- AXIS Clinicals Limited, Miyāpur, Hyderabad, India